CLINICAL TRIAL: NCT03124134
Title: A Randomized, Open-label, Crossover Study Assessing the Effects of Gelesis200 on Glucose and Insulin Following a Single Administration of Gelesis200 in Healthy Subjects
Brief Title: Gelesis Glycemic Index Study
Acronym: GLIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gelesis, Inc. (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GS-200-005; 160159 (Other: inVentiv Health Clinique)
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Obesity; Diabetes; PreDiabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Prediabetic State | interventions — Water; Single Person

STUDY DESIGN:
Intervention Model Description: 4-way crossover with the option for 2 more crossover arms after interim analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- A) Gelesis200, 50 g carbs (Experimental): 4.20 g of Gelesis200 before a 50 g carbohydrate breakfast
  Interventions: Device: Gelesis200
- B) Gelesis200, 100 g carbs (Experimental): 4.20 g of Gelesis200 before a 100 g carbohydrate breakfast
  Interventions: Device: Gelesis200
- C) Water, 50 g carbs (Placebo Comparator): 300 mL water before a 50 g carbohydrate breakfast
  Interventions: Other: Water, only (placebo)
- D) Water, 100 g carbs (Placebo Comparator): 300 mL water before a 100 g carbohydrate breakfast
  Interventions: Other: Water, only (placebo)
- E) Gelesis200, TBD carbs (Experimental): up to 4.20 g Gelesis200 before a meal of either 50 g or 100 g carbohydrate breakfast (to be determined after interim analysis)
  Interventions: Device: Gelesis200
- F) Water, TBD carbs (Placebo Comparator): 300 mL of water before a meal of either 50 g or 100 g carbohydrate breakfast (to be determined after interim analysis)
  Interventions: Other: Water, only (placebo)

INTERVENTIONS:
Device: Gelesis200 — Encapsulated hydrogel
  Arms: A) Gelesis200, 50 g carbs; B) Gelesis200, 100 g carbs; E) Gelesis200, TBD carbs
Other: Water, only (placebo) — 300 mL of water
  Arms: C) Water, 50 g carbs; D) Water, 100 g carbs; F) Water, TBD carbs

SUMMARY:
A study to determine glucose and insulin responses to 50g and 100 g of carbohydrate with and without Gelesis200.

DETAILED DESCRIPTION:
This will be a single centre, open-label, randomized, single-administration, 4-period, 4-way, crossover, pilot study with glycemic and insulin assessments. There is also an option for 2 additional single-administration periods based on the results of an interim analysis.

The study includes 2 treatments arms with Gelesis200 (4.20 g 10 minutes before a 50 g carbohydrate breakfast and 4.20 g 10 minutes before a 100 g carbohydrate breakfast) plus 2 control arms consisting of consumption of the breakfasts with water only.

The optional periods consist of 1 treatment arm with Gelesis200 and 1 control arm with breakfast and water only. Either only one or both the optional periods may be conducted. The number of additional period(s) to conduct, the amount of Gelesis200 in the treatment arm, as well as the meal composition will be based on interim analysis results.

ELIGIBILITY:
Inclusion Criteria:

1. Male.
2. Non-smoker (no use of tobacco products within 6 months prior to screening), ≥ 22 and ≤ 65 years of age, with body mass index (BMI) ≥ 18.5 and < 30.0 kg/m2.
3. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 12 weeks prior to administration. Subjects vomiting within 24 hours pre-administration will be carefully evaluated for upcoming illness/disease. Inclusion pre-administration is at the discretion of the Qualified Investigator.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease, including, but not limited to pancreatitis, hepatitis B or C, HIV, swallowing disorders, and gastroesophageal reflux disease (at least 1 episode per week).
   3. the absence of clinically significant history of gastric or peptic ulcer, small bowel resection (except if related to appendectomy), intestinal stricture (e.g., Crohn's disease), intestinal obstruction or high risk of intestinal obstruction including suspected small bowel adhesions.
   4. the absence of clinically significant history or known presence of esophageal anatomic abnormalities (e.g., webs, diverticuli, rings), gastroparesis, and malabsorption.
   5. the absence of history of gastric bypass, any other gastric surgery and intragastric balloon.
   6. the absence of history of angina, coronary bypass, and myocardial infarction within 6 months prior to administration.
   7. the absence of history of abdominal radiation treatment.
   8. the absence of history of cancer within the past 5 years, except adequately-treated localized basal cell skin cancer.
4. Capable of consent.
5. Fasting plasma glucose < 100 mg/dL (< 5.6 mmol/L) and fasting insulin < 10 μIU/mL (< 69.5 pmol/L) at screening.
6. Ability and willingness to consume 3 slices of white bread within 10 minutes and 6 slices of white bread within 15 minutes.

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen at screening.
3. History of allergic reactions to carboxymethylcellulose, citric acid, gelatin, titanium dioxide, or other related substances.
4. Any reason which, in the opinion of the Qualified Investigator, would prevent the subject from participating in the study.
5. Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
6. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
7. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
8. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first IP administration, administration of a biological product in the context of a clinical research study within 90 days prior to the first IP administration, or concomitant participation in an investigational study involving no drug or device administration.
9. Use of medication other than topical products without significant systemic absorption:

   1. prescription medication within 30 days prior to the first administration;
   2. over-the-counter products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first administration, with the exception of the occasional use of acetaminophen (up to 2 g daily);
   3. a depot injection or an implant of any drug within 3 months prior to the first administration.
10. Donation of plasma within 7 days prior to administration. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL within 30 days, or more than 499 mL within 56 days prior to the first administration.
11. Hemoglobin < 128 g/L and hematocrit < 0.37 L/L at screening.
12. Glycosylated hemoglobin (HbA1c) ≥ 6.5% (≥ 48 mmol/mol) at screening.
13. Serum low-density lipoprotein cholesterol ≥ 190 mg/dL (≥ 4.93 mmol/L) at screening.
14. Serum triglycerides ≥ 500 mg/dL (≥ 5.65 mmol/L) at screening.
15. Abnormal TSH at screening, or abnormal free T4 if TSH is slightly out of range.
16. Anticipating surgical intervention during the study.

Ages: 22 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | single administration on each of up to 6 days over 6 weeks
  AEs, lab abnormalities

SECONDARY OUTCOMES:
Post prandial glucose | single administration on each of up to 6 days over 6 weeks
  iAUC of glucose after a carbohydrate containing meal
Post prandial insulin | single administration on each of up to 6 days over 6 weeks
  iAUC of insulin after a carbohydrate containing meal

CONTACTS AND LOCATIONS:
Overall Officials: Audet, Principal Investigator — inVentiv Health Clinique
Locations (1):
- inVentiv Health Clinique, Québec, Canada

IPD SHARING:
Plan to Share IPD: No
The individual data will not be available to other researchers.